CLINICAL TRIAL: NCT01665560
Title: Neural, Behavioral and Physiological Correlates of Feeding in Humans
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0505027690
Record Dates: First submitted 2012-08-02; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Magnetic Resonance Imaging, Functional
Keywords: smoking; fMRI; odors; taste
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva samples were obtained and are stored using a coded ID in a secure part of our facility
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Smokers--Currently Smoking: Individuals that are right handed, and not claustrophobic were recruited. This same group was used for the smoking-group and refrain from smoking was evaluated by CO2 evaluation. To be classified as smokers, they had to report smoking 3-10 cigarettes daily for at least the last year and have a carbon monoxide reading of CO >10 ppm.
- Non-Smoker: Healthy individuals meeting the inclusion criteria who claim to not smoke. This is confirmed w/ CO testing.

SUMMARY:
The overarching goal of this project is to understand how nicotine addiction interacts with feeding behaviors and brain representation of food reward. The current proposal is part of a larger effort to begin a program of research to elucidate similarities and differences in perception of, and behavioral and neural response to, food and cigarette aromas as a function of 1) smoking status (smokers, ex-smokers who do gain weight, ex-smokers who do not gain weight, non-smokers), 2) internal state (hungry, full), and 3) cigarette deprivation (acute, chronic). A general hypothesis is that there are overlapping neural mechanisms governing food reward and cigarette reward in smokers and that this overlap includes incentive salience encoding.

DETAILED DESCRIPTION:
Weight gain frequently follows smoking cessation. Fear of weight gain is cited as a key reason not to quit and actual weight gain is a primary reason for relapse, especially among women. Although the causes of weight gain following smoking cessation are complex, increased caloric intake is recognized as one of the primary sources. One explanation for increased caloric intake is that, there are common neural mechanisms for food and cigarette reward and hence food reward can substitute for cigarette reward and vice versa. An alternative explanation for weight gain following smoking cessation is that there is an overall decrease in brain reward function during nicotine withdrawal, which leads to a decrease in the reward value of food and consequent increase in intake to maintain the total amount of reward obtained by food. The success of the proposed studies relies upon our ability to deliver odorants in the fMRI scanner and to measure neural activation in regions such as the amygdala, which are susceptible to inhomogeneity artifacts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* between the ages of 18-45
* fMRI safe

Exclusion Criteria:

* outside of the above age range
* not able to have an fMRI (non-removable metal, pacemaker, etc)
* medical diagnosis related to neurological problems, anxiety, psychiatric conditions
* Did not refrain from smoking for the described time in the smoking group, or showed a CO2 level consistent with a smoker in the non-smoking group

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults in the New Haven, CT area.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2005-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
fMRI w/ taste and smell stimuli | 1-2 hours
  Subjects will be scanned on a 3T Trio magnet while tasting and smelling various food and non-food substances. Our primary outcome measure will be differential brain responses to taste and smell stimuli as a function of group (smokers vs. nonsmokers).

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Small, PhD, Principal Investigator — Yale & John B Pierce Laboratory
Locations (1):
- John B Pierce Laboratory, New Haven, Connecticut, United States